CLINICAL TRIAL: NCT04469478
Title: The Use of Virtual Reality for Diagnostic Imaging Review With Cancer Patients
Brief Title: Virtual Reality in Imaging Review for Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not approved in 2020 secondary to COVID-19 restrictions on trials
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0560.cc
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Patient Education; Virtual Reality; Diagnostic Imaging; Cancer Patient
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Single Arm Exploratory Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality for imaging review (Experimental): Each participant (patient and caregiver(s)) will undergo standard 2D imaging review on a computer screen, followed by 3D imaging review in virtual reality during their radiation oncology consultation
  Interventions: Other: Survey and interview

INTERVENTIONS:
Other: Survey and interview — Patients and caregivers will provide information via surveys and interviews regarding their experience viewing diagnostic imaging using conventional methods and using Virtual Reality

SUMMARY:
Patients with cancer and their caregivers may have difficulty understanding the site and extent of their disease. Poor comprehension may negatively impact patients and caregivers, leading to increased anxiety, reduced compliance, decreased trust of the physician, and limited shared medical decision making ability. Most patients want to be thoroughly informed, with over a third of cancer patients wishing they had been better informed about side effects that they experienced due to their treatment. The purpose of this study is to evaluate the impact of diagnostic imaging review using 3D virtual reality compared to standard 2D imaging review for patients and their caregiver(s) using a mixed methods approach of survey and qualitative interview based approaches.

DETAILED DESCRIPTION:
This study will use virtual reality to display the patient's diagnostic imaging in 3D with live volumetric rendering. This study will explore if this approach improves patient and caregiver understanding of their disease. Eligible patients should have available diagnostic imaging consisting of CT, MRI, and/or PET-CT. Prior to their consultation in radiation oncology, patients will complete a survey about their prior experience reviewing their diagnostic imaging. During the consultation, patients and caregivers will be shown their medical imaging in 2D on a computer screen, then in 3D with virtual reality. After the consultation, the patient and caregiver(s) will complete a 2nd survey comparing virtual reality to standard imaging review with domains of perceived understanding, patient preference, and satisfaction. Then, the patient and caregiver(s) will undergo a qualitative interview exploring their experience with virtual reality compared to standard imaging review. The survey questions comparing virtual reality to standard imaging review will be statistically evaluated. The recorded interview session will be qualitatively analyzed using with a mixed methods approach by thematically categorizing the respondents' answers.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign and date the consent form.
* Willingness to comply with all study procedures and be available for the duration of the study.
* Male or female patient 18 years or older.
* Available diagnostic imaging (MRI, CT and/or PET)
* Consultation in radiation oncology for consideration of radiation therapy.
* English speaking.

Exclusion Criteria:

* Inability to complete virtual reality, survey and interview.
* Non-English speaking
* Patients with visual defects that affect their ability to view content in VR

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Successful Completion of Imaging Review Using Virtual Reality | During the consultation 1 day visit
  The percentage of patients able to complete the review of their imaging using virtual reality

SECONDARY OUTCOMES:
Satisfaction and preference | During the consultation 1 day visit
  Evaluate patients' and caregivers' satisfaction and preferences regarding diagnostic imaging review using a focused survey
Qualitative feedback regarding imaging review using virtual reality | During the consultation 1 day visit
  Collect patients' and caregivers' feedback regarding imaging review using virtual reality through qualitative interviews.
Baseline demographics and imaging review experience | During the consultation 1 day visit
  Capture baseline demographics, education, and prior experience with diagnostic imaging review.
Intervention time interval | During the consultation 1 day visit
  Measure the time spent reviewing diagnostic imaging with virtual reality and standard approaches relative to the consultation time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Anschutz Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernsler JI, Cannon CA. The whys of patient education. Semin Oncol Nurs. 1991 May;7(2):79-86. doi: 10.1016/0749-2081(91)90085-4. PMID 1882153
- [Background] Gold DT, McClung B. Approaches to patient education: emphasizing the long-term value of compliance and persistence. Am J Med. 2006 Apr;119(4 Suppl 1):S32-7. doi: 10.1016/j.amjmed.2005.12.021. PMID 16563940
- [Background] Hess CB, Chen AM. Measuring psychosocial functioning in the radiation oncology clinic: a systematic review. Psychooncology. 2014 Aug;23(8):841-54. doi: 10.1002/pon.3521. Epub 2014 May 21. PMID 24846702
- [Background] Takahashi T, Hondo M, Nishimura K, Kitani A, Yamano T, Yanagita H, Osada H, Shinbo M, Honda N. Evaluation of quality of life and psychological response in cancer patients treated with radiotherapy. Radiat Med. 2008 Aug;26(7):396-401. doi: 10.1007/s11604-008-0248-5. Epub 2008 Sep 4. PMID 18769996
- [Background] Johnson A, Sandford J. Written and verbal information versus verbal information only for patients being discharged from acute hospital settings to home: systematic review. Health Educ Res. 2005 Aug;20(4):423-9. doi: 10.1093/her/cyg141. Epub 2004 Nov 30. PMID 15572437
- [Background] Theis SL, Johnson JH. Strategies for teaching patients: a meta-analysis. Clin Nurse Spec. 1995 Mar;9(2):100-5, 120. doi: 10.1097/00002800-199503000-00010. PMID 7600475
- [Background] Friedman AJ, Cosby R, Boyko S, Hatton-Bauer J, Turnbull G. Effective teaching strategies and methods of delivery for patient education: a systematic review and practice guideline recommendations. J Cancer Educ. 2011 Mar;26(1):12-21. doi: 10.1007/s13187-010-0183-x. PMID 21161465
- [Background] Press Ganey: public reporting gives huge boost to patient satisfaction. Healthcare Benchmarks Qual Improv. 2008 Dec;15(12):121-3. PMID 19024286
- [Background] Meredith C, Symonds P, Webster L, Lamont D, Pyper E, Gillis CR, Fallowfield L. Information needs of cancer patients in west Scotland: cross sectional survey of patients' views. BMJ. 1996 Sep 21;313(7059):724-6. doi: 10.1136/bmj.313.7059.724. PMID 8819442
- [Background] Shaverdian N, Yeboa DN, Gardner L, Harari PM, Liao K, McCloskey S, Tuli R, Vapiwala N, Jagsi R. Nationwide Survey of Patients' Perspectives Regarding Their Radiation and Multidisciplinary Cancer Treatment Experiences. J Oncol Pract. 2019 Dec;15(12):e1010-e1017. doi: 10.1200/JOP.19.00376. Epub 2019 Nov 20. PMID 31747336